CLINICAL TRIAL: NCT01005511
Title: A Single Centre, Randomised, Clinical Placebo Controlled Study of the Optimal Treatment and Long-term Effect of FES on Sleep Bruxism
Brief Title: Treatment Period and Long-term Efficacy of Functional Electrical Stimulation (FES) on Sleep Bruxism
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: The population described via ex- and inclusion criteria did not excisit
Sponsor: Medotech A/S (Industry)
Responsible Party: Peter Svensson, Aarhus University Dentist School
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: TMD-01
Record Dates: First submitted 2009-10-30; First posted 2009-11-02 (Estimated); Last update posted 2011-06-08 (Estimated); Status verified 2009-10

CONDITIONS: Bruxism
Keywords: Bruxism
MeSH Terms: conditions — Bruxism

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Grindcare (Experimental): 24 patients receiving active treatment
  Interventions: Device: Grindcare
- Placebo treatment (Placebo Comparator): 24 patients receive a placebo treatment
  Interventions: Device: Grindcare - inactive

INTERVENTIONS:
Device: Grindcare — Active treatment
  Arms: Grindcare
Device: Grindcare - inactive — Placebo treatment
  Arms: Placebo treatment

SUMMARY:
To investigate the effect of the treatment with Grindcare® on the muscles- and jaw symptoms and at the jaw muscle activity during sleep.

ELIGIBILITY:
Inclusion Criteria:

* Signed and dated ICF
* 18 years or older
* Fulfill the RDC-criteria for myofascial TMD diagnose (group 1a or 1b)

Exclusion Criteria:

* Contraindication of concommitant diseases for the study judged by investigator
* Patients who are using occlusal splints in the treatment period.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Estimated)
Dates: Start 2009-10; Primary Completion 2010-10 (Actual); Study Completion 2010-12 (Actual)

PRIMARY OUTCOMES:
Reduction in the electromyography (EMG) activity per hour per night | 10 weeks after start of treatment

SECONDARY OUTCOMES:
Evaluation of long-term effect of FES on the EMG activity | a 4 weeks period after end og treatment with FES

CONTACTS AND LOCATIONS:
Overall Officials: pernille Wendelboe, MsSc (Odont), Study Chair — Medotech A/S
Locations (1):
- Odontologisk Institute, Aarhus, Denmark